CLINICAL TRIAL: NCT00818350
Title: Phase II Study of Sunitinib in Metastatic and Pretreated Urothelial Cancer
Brief Title: Activity Study of Sunitinib In Metastatic Pretreated Urothelial Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Campania Younger Oncologists Association (Other)
Responsible Party: DI LORENZO GIUSEPPE, AGOC
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AGOC O1
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- SUNITINIB (Experimental)
  Interventions: Drug: SUNITINIB

INTERVENTIONS:
Drug: SUNITINIB — 50 MG ORAL, DAYS 1-28 FOLLOWED BY 2 WEEKS RESTING
  Other Names: SUTENT

SUMMARY:
Gemcitabine and cisplatin represent the standard first-line chemotherapy in metastatic bladder carcinoma. This regimen has replaced in most centers the MVAC combination showing a similar efficacy but less toxicity.

Almost all responding patients relapse within the first year, with a median survival of 12 months. Prognosis is very poor in patients who display progressive disease after receiving combination cisplatin-based chemotherapy.

No standard has yet been established for second-line treatment and well designed trials of second-line chemotherapy for metastatic transitional carcinoma of the urothelium should be given high priority.

Several drugs have been used in second line for metastatic disease with poor results.

The investigators have planned a Phase II study, open-label, single arm design to evaluate the activity and safety of sunitinib in metastatic urothelial carcinoma, pretreated with standard regimen (cisplatin-gemcitabine).

No previous studies have been published with sunitinib in metastatic bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES

* PRIMARY To determine the antitumor efficacy ( response rate) of sunitinib
* SECONDARY To determine: safety, duration of response, Quality of life (QoL), progression free survival (PFS) and overall survival (OS).

PLAN OF TREATMENT Patients received sunitinib at a starting dose of 50 mg per day in repeated 6-week cycles for 4 consecutive weeks followed by 2 weeks off treatment.

Sunitinib was self-administered orally once daily without regard to meals. Dose reduction for toxicity was allowed to 37.5 until 25 mg/day depending on the type and severity of toxicity encountered.

Sunitinib treatment was continued until disease progression, unacceptable toxicity or withdrawal of consent.

EVALUATION

Baseline evaluations included:

* medical history
* physical examination;
* tumor assessment (total body TC and bone scan )
* assessment of ECOG PS
* QoL assessment
* Assessment of left ventricular ejection fraction by echocardiography
* ECG
* Laboratory measurements. Assessment of efficacy and safety
* Evaluation according RECIST criteria every 2 cycles (12 weeks) with TC
* Safety according NCI version 3 every cycle
* QoL every cycle EORTC-QOL-C30.• RESOURCE UTILIZATION ASSESSMENTS

EORTC QLQ-C30 questionnaire, developed by the EORTC for the measurement of quality of life in cancer patients in clinical trials.

For the analysis, the raw scores of the questionnaire are transformed into a 100-point scale. For the functional scales, the computed scores range from 0 to 100, with the higher scores representing a higher level of functioning. For the item scales relative to physical symptoms and financial impact, higher scores represent a higher level of symptoms or problems .

STATISTICAL METHODS

Benefit anticipated (%): >30% of response rate. Test size: 5%. Power 80%. Sample size: 25 patients.

ELIGIBILITY:
Inclusion Criteria:

* cytological confirmation of UROTHELIAL carcinoma
* Failure of Cisplatin-gemcitabine regimen as first-line
* Presence of measurable metastases
* Performance status 0-1 ECOG
* Age of 18 years or older
* Written informed consent
* Adequate organ function ( based on tests of hematologic, hepatic, renal and cardiac function).

Exclusion Criteria:

* administration of a previous biological therapy ( sorafenib , bevacizumab or mTor Inhibitor)
* brain metastases
* significant cardiac events within the 6 months prior to study drug administration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
To determine the antitumor efficacy ( response rate) of sunitinib | 12 weeks

SECONDARY OUTCOMES:
QOL | 6 WEEKS
TOXICITY ACCORDING NCI VERSION 3 CRITERIA | EVERY WEEK

CONTACTS AND LOCATIONS:
Overall Officials: DI LORENZO GIUSEPPE, PHD, Principal Investigator — Campania Younger Oncologists Association